CLINICAL TRIAL: NCT06308081
Title: SMART: Social Media Anti-Vaping Messages to Reduce ENDS Use Among Sexual and Gender Minority Teens
Brief Title: Social Media Anti-Vaping Messages to Reduce ENDS Use Among Sexual and Gender Minority Teens
Acronym: SMART
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Abramson Cancer Center at Penn Medicine (Other)
Collaborators: University of Florida (Other)
Responsible Party: Principal Investigator, Andy Tan, Associate Professor of Communication, Abramson Cancer Center at Penn Medicine
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: UPCC 13023; 849052 (Other: University of Pennsylvania)
Record Dates: First submitted 2024-01-03; First posted 2024-03-13 (Actual); Last update posted 2025-10-07 (Actual); Status verified 2025-10

CONDITIONS: Vaping; Adolescent Behavior; Communication Research
Keywords: Communication interventions; LGBTQ+ youth
MeSH Terms: conditions — Vaping; Adolescent Behavior

STUDY DESIGN:
Intervention Model Description: Participants will be randomized to 1 of 2 conditions: SGM-tailored anti-vaping messages versus non-tailored messages. Block randomization will achieve balance across the two conditions based on age group, gender identity, sexual orientation, race, ethnicity, and prior use. Both conditions will receive repeated exposure of messages within their assigned condition daily for 4, up to a total of 24 messages over the course of the study. Messages will be delivered using texting to participants mobile phones. We will record participants' self-reported engagement to the messages at the follow-up survey (after measuring the study outcomes). Participants will be asked to complete a baseline survey comprising vaping susceptibility and characteristics, surveys at 1-, 2-, 3-, and 4-weeks follow-up to measure vaping susceptibility.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Tailored (Experimental): Participants in the tailored arm will receive SGM-tailored anti-vaping health messages delivered via text message
  Interventions: Other: Tailored
- Non-Tailored (No Intervention): Participants in the non-tailored arm will receive non-tailored anti-vaping health messages delivered via text message

INTERVENTIONS:
Other: Tailored — Messages will be in the form of high-quality English-language anti-vaping messages comprising static text and imagery designed to resemble social media posts (e.g., image and a caption). We will create 24 messages based on the top-ranked tailoring features and belief themes tested in Aim 2 to comprise SGM-tailored messages. For the non-tailored message condition, we will create 24 anti-vaping social media messages that mirror the SGM-tailored messages but do not contain SGM identity cues. We will match the belief themes used in the tailored and non-tailored messages such that they represent a range of belief targets (e.g., addiction, physical health effects, mental health effects) as indicated in Aims 1 and 2. We do not utilize a social media platform for the delivery of the message to avoid potential contamination across randomized conditions.
  Other Names: SGM tailored messages
  Arms: Tailored

SUMMARY:
The investigators long-term goal is to reduce tobacco use and tobacco-related health disparities among SGM populations. The objective of Project SMART (Social Media Anti-Vaping Messages to Reduce ENDS Use Among Sexual and Gender Minority Teens) is to evaluate the effectiveness of an sexual gender minority (SGM) -tailored social media intervention to prevent vaping initiation among SGM youth ages 13-20 years. The investigators central hypothesis is that SGM-tailored anti-vaping social media messages will be more effective than existing non-tailored messages to prevent vaping initiation among SGM youth. The scientific premise for this work is based on principles of cultural tailoring in health communication for vulnerable populations, the Health Equity Promotion Model, and the Message Impact Framework. The investigators are developing and evaluating a social media intervention because SGM youth have a high rate of social media use and are more likely to go online for health information than non-SGM youth. Social media, moreover, are increasingly used for health promotion to address health disparities and well-being of SGM populations. The investigators will conduct rapid-cycle feedback with stakeholders including SGM organization leaders to provide input on the message design, testing, and intervention implementation to ensure feasibility and acceptability of the intervention.

DETAILED DESCRIPTION:
Aim 1: Explore salient beliefs and cultural tailoring preferences related to vaping initiation among sexual gender minority (SGM) youth to inform the development of anti-vaping social media messages.

Approach: An elicitation survey among 80 SGM youth and focus group discussions among a subsample of 48-64 youth who complete the elicitation survey will explore beliefs related to vaping initiation that SGM youth find most salient. Participants will include US SGM youth, ages 12-18 years, stratified by age (12-15 or 16-18), vaping status (never vaped and are susceptible or have initiated vaping in the past 1 year), and gender identity (cisgender or transgender/gender expansive). The investigators will further explore the social contexts of their vaping behavior and preferences for cultural tailoring of anti-vaping messages (i.e., peripheral, evidential, linguistic, and sociocultural values tailoring) among SGM youth.

Aim 2: Identify promising anti-vaping social media messages and cultural tailoring strategies to reduce vaping initiation among SGM youth.

Approach: Results from Aim 1 and input from community stakeholders will be utilized to develop SGM-tailored social media anti-vaping messages. An online discrete choice experiment among SGM youth ages 13-18 years (n=600) who have never vaped will be used to test the impact of anti-vaping messages and cultural tailoring strategies on perceived message effectiveness to reduce vaping initiation. Results will guide the construction of culturally tailored anti-vaping social media intervention for broader evaluation in Aim 3.

Aim 3: Evaluate the effectiveness of repeated exposure to SGM-tailored anti-vaping social media messages on subsequent vaping susceptibility among SGM youth.

Approach: The investigators will conduct a prospective 2-group randomized experiment among 1500 SGM youth and young adults ages 13-20 to test the hypothesis that repeated exposure to SGM-tailored anti-vaping social media messages will be associated with reduced vaping susceptibility, defined as the extent to which youth are open to vaping, compared with non-tailored messages.

ELIGIBILITY:
Inclusion Criteria:

* Identify as SGM
* ages 13-20
* not vaped or used other tobacco products in the past 30 days
* have access to a smartphone
* Able to read and speak in English
* willing to receive messages via texting for the study
* susceptible to e-cigarette use at intake (i.e., those do not state "definitely not" to all three susceptibility questions).

Exclusion Criteria:

* Current vapers
* Non-SGM youth

Ages: 13 Years to 20 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 1155 (Actual)
Dates: Start 2024-02-21 (Actual); Primary Completion 2025-08-15 (Actual); Study Completion 2025-08-15 (Actual)

PRIMARY OUTCOMES:
Susceptibility to vaping | One week, Two weeks, Three weeks, and One month
  We will measure susceptibility to vaping using four items previously used on PATH Wave 7 youth questionnaire and NYTS 2022 Questionnaire:
  1. Have you ever been curious about using an e-cigarette or other electronic nicotine products? (1 = Not at all curious; 2 = A little curious; 3 = Somewhat curious; 4 = Very curious)
  2. Do you think you will use an e-cigarette or an electronic nicotine product in the next year? (1 = Definitely not; 2 = Probably not; 3 = Probably yes; 4 = Definitely yes)
  3. Do you think you will use an e-cigarette or an electronic nicotine product soon? (1 = Definitely not; 2 = Probably not; 3 = Probably yes; 4 = Definitely yes)
  4. If one of your best friends were to offer you an e-cigarette or an electronic nicotine product, would you use it? (1 = Definitely not; 2 = Probably not; 3 = Probably yes; 4 = Definitely yes)
  The responses to these items will be averaged to create a score of vaping susceptibility.

SECONDARY OUTCOMES:
Vaping initiation | One week, Two weeks, Three weeks, and One month
  We will measure vaping initiation in the past 1 week using one item:
  1) Have you used an e-cigarette or vape, even once or twice in the past week? (1 = Yes; 2 = No)

CONTACTS AND LOCATIONS:
Locations (1):
- University of Pennsylvania, Philadelphia, Pennsylvania, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Bold KW, Kong G, Cavallo DA, Camenga DR, Krishnan-Sarin S. E-Cigarette Susceptibility as a Predictor of Youth Initiation of E-Cigarettes. Nicotine Tob Res. 2017 Dec 13;20(1):140-144. doi: 10.1093/ntr/ntw393. PMID 28035000
- [Background] Seo DC, Kwon E, Lee S, Seo J. Using susceptibility measures to prospectively predict ever use of electronic cigarettes among adolescents. Prev Med. 2020 Jan;130:105896. doi: 10.1016/j.ypmed.2019.105896. Epub 2019 Nov 12. PMID 31730945
- [Background] Noar SM, Gottfredson NC, Kieu T, Rohde JA, Hall MG, Ma H, Fendinger NJ, Brewer NT. Impact of Vaping Prevention Advertisements on US Adolescents: A Randomized Clinical Trial. JAMA Netw Open. 2022 Oct 3;5(10):e2236370. doi: 10.1001/jamanetworkopen.2022.36370. PMID 36227597
- [Background] Kasza KA, Edwards KC, Tang Z, Stanton CA, Sharma E, Halenar MJ, Taylor KA, Donaldson E, Hull LC, Day H, Bansal-Travers M, Limpert J, Zandberg I, Gardner LD, Hammad HT, Borek N, Kimmel HL, Compton WM, Hyland A. Correlates of tobacco product initiation among youth and adults in the USA: findings from the PATH Study Waves 1-3 (2013-2016). Tob Control. 2020 May;29(Suppl 3):s191-s202. doi: 10.1136/tobaccocontrol-2020-055671. PMID 32321853
- [Background] Stanton CA, Sharma E, Seaman EL, Kasza KA, Edwards KC, Halenar MJ, Taylor KA, Day H, Anic G, Hull LC, Bansal-Travers M, Limpert J, Gardner LD, Hammad HT, Borek N, Kimmel HL, Compton WM, Hyland A. Initiation of any tobacco and five tobacco products across 3 years among youth, young adults and adults in the USA: findings from the PATH Study Waves 1-3 (2013-2016). Tob Control. 2020 May;29(Suppl 3):s178-s190. doi: 10.1136/tobaccocontrol-2019-055573. PMID 32321852
- [Background] Kushins L. Clonidine withdrawal, propranolol, and rebound hypertension. Anesthesiology. 1980 Aug;53(2):178-9. doi: 10.1097/00000542-198008000-00017. No abstract available. PMID 7416532
- [Background] Neer CS 2nd, Grantham SA, Foster RR. Femoral shaft fracture with sciatic nerve palsy. JAMA. 1970 Dec 28;214(13):2307-11. No abstract available. PMID 5537073
- [Background] Lazard AJ. Social Media Message Designs to Educate Adolescents About E-Cigarettes. J Adolesc Health. 2021 Jan;68(1):130-137. doi: 10.1016/j.jadohealth.2020.05.030. Epub 2020 Jul 9. PMID 32654836
- [Background] Ossenberg FW, Martin W, Saegler J, Haan D. [Changes in enzyme activities during poisoning]. Cah Med. 1970 Oct 30;11(12):1055-9. No abstract available. French. PMID 5485217
- [Background] Tabaac AR, Haneuse S, Johns M, Tan ASL, Austin SB, Potter J, Lindberg L, Charlton BM. Sexual and reproductive health information: Disparities across sexual orientation groups in two cohorts of U.S. women. Sex Res Social Policy. 2021 Sep;18(3):612-620. doi: 10.1007/s13178-020-00485-3. Epub 2020 Jul 22. PMID 34484460
- [Background] Lang S, Bantic Z, Jakupcevic M, Sosic Z, Mitak M, Nasic M. [Medical ethics in the curriculum of the School of Medicine at the University in Zagreb]. Lijec Vjesn. 1984 Jan;106(1):39-42. No abstract available. Croatian. PMID 6708717
- [Background] Katz-Wise SL, Ehrensaft D, Vetters R, Forcier M, Austin SB. Family Functioning and Mental Health of Transgender and Gender-Nonconforming Youth in the Trans Teen and Family Narratives Project. J Sex Res. 2018 May-Jun;55(4-5):582-590. doi: 10.1080/00224499.2017.1415291. Epub 2018 Jan 16. PMID 29336604
- [Background] Sachs BA, Wolfman L, Herzig N. Plasma lipid and lipoprotein alterations during oral contraceptive administration. Obstet Gynecol. 1969 Oct;34(4):530-5. No abstract available. PMID 5822679
- [Background] Dupont C, Ciaburro H, Prevost Y, Cloutier G. Phenol skin tightening for better dermabrasion. Plast Reconstr Surg. 1972 Dec;50(6):588-90. doi: 10.1097/00006534-197212000-00007. No abstract available. PMID 4636492
- [Background] Fishbein M, Ajzen I. Predicting and changing behavior: the reasoned action approach. New York: Psychology Press; 2010.
- [Background] Bates SR, Murphy PL, Feng ZC, Kanazawa T, Getz GS. Very low density lipoproteins promote triglyceride accumulation in macrophages. Arteriosclerosis. 1984 Mar-Apr;4(2):103-14. doi: 10.1161/01.atv.4.2.103. PMID 6704048
- [Background] Szymanski DM. Does Internalized Heterosexism Moderate the Link Between Heterosexist Events and Lesbians' Psychological Distress? Sex Roles. 2006 Feb 1;54(3-4):227-234.
- [Background] Testa RJ, Habarth J, Peta J, Balsam K, Bockting W. Development of the Gender Minority Stress and Resilience Measure. Psychology of Sexual Orientation and Gender Diversity. US: Educational Publishing Foundation; 2015;2(1):65-77.
- [Background] Meyer IH, Rossano L, Ellis JM, Bradford J. A brief telephone interview to identify lesbian and bisexual women in random digit dialing sampling. J Sex Res. 2002 May;39(2):139-44. doi: 10.1080/00224490209552133. PMID 12476246
- [Background] Smith BW, Dalen J, Wiggins K, Tooley E, Christopher P, Bernard J. The brief resilience scale: assessing the ability to bounce back. Int J Behav Med. 2008;15(3):194-200. doi: 10.1080/10705500802222972. PMID 18696313
- [Background] Foulds J, Veldheer S, Yingst J, Hrabovsky S, Wilson SJ, Nichols TT, Eissenberg T. Development of a questionnaire for assessing dependence on electronic cigarettes among a large sample of ex-smoking E-cigarette users. Nicotine Tob Res. 2015 Feb;17(2):186-92. doi: 10.1093/ntr/ntu204. Epub 2014 Oct 19. PMID 25332459
- [Background] Centers for Disease Control and Prevention, National Center for Chronic Disease Prevention and Health Promotion, Division of Population Health. CDC BRFSS Questionnaires [Internet]. 2018 [cited 2018 May 14]. Available from: https://www.cdc.gov/brfss/questionnaires/index.htm
- [Background] Moir DD, Willocks J. Continuous epidural analgesia in inco-ordinate uterine action. Acta Anaesthesiol Scand Suppl. 1966;23:144-53. doi: 10.1111/j.1399-6576.1966.tb01005.x. No abstract available. PMID 5304983
- [Background] Doxbeck CR. Up in Smoke: Exploring the Relationship between Bullying Victimization and E-Cigarette Use in Sexual Minority Youths. Subst Use Misuse. 2020;55(13):2221-2229. doi: 10.1080/10826084.2020.1797809. Epub 2020 Jul 28. PMID 32720554
- [Background] Lanzieri CF, Duchesneau PM, Rosenbloom SA, Smith AS, Rosenbaum AE. The significance of asymmetry of the foramen of Vesalius. AJNR Am J Neuroradiol. 1988 Nov-Dec;9(6):1201-4. PMID 3143245
- [Background] Johns MM, Pingel ES, Youatt EJ, Soler JH, McClelland SI, Bauermeister JA. LGBT community, social network characteristics, and smoking behaviors in young sexual minority women. Am J Community Psychol. 2013 Sep;52(1-2):141-54. doi: 10.1007/s10464-013-9584-4. PMID 23783884
- [Background] Via'lba EV, Iushchuk ND, Belaia IuA. [Detection of Yersinia antigens in biological substrates from adult patients with Yersinia infection]. Sov Med. 1989;(4):96-7. No abstract available. Russian. PMID 2762930
- [Background] Rideout V, Robb MB. Social media, social life: Teens reveal their experiences [Internet]. San Francisco, CA: Common Sense Media; 2018. Available from: https://www.commonsensemedia.org/sites/default/files/uploads/research/2018_cs_socialmediasociallife_fullreport-final-release_2_lowres.pdf
- [Background] Mielens ZE, Drobeck HP, Rozitis J Jr, Sansone VJ Jr. Interaction of aspirin with nonsteroidal anti-inflammatory drugs in rats. J Pharm Pharmacol. 1968 Jul;20(7):567-9. doi: 10.1111/j.2042-7158.1968.tb09807.x. No abstract available. PMID 4386615
- [Background] Hatzenbuehler ML, Wieringa NF, Keyes KM. Community-level determinants of tobacco use disparities in lesbian, gay, and bisexual youth: results from a population-based study. Arch Pediatr Adolesc Med. 2011 Jun;165(6):527-32. doi: 10.1001/archpediatrics.2011.64. PMID 21646585
- [Background] Formaziuk VE, Dobretsov GE, Deev AI, Vladimirov IuA. [Estimation of the density of the surface charge in lipoproteins from human blood plasma]. Vopr Med Khim. 1982 Jan-Feb;28(1):119-22. No abstract available. Russian. PMID 7064376
- [Background] Igboeli G, Rakha AM. Bull testicular and epididymal functions after long-term vasectomy. J Anim Sci. 1970 Jul;31(1):72-5. doi: 10.2527/jas1970.31172x. No abstract available. PMID 4915974
- [Background] Trebukhin MV. [Use of hexachlorparaxylol in fascioliasis]. Veterinariia. 1971 Aug;9:68-9. No abstract available. Russian. PMID 5140682
- [Background] Iwata F, Joh T, Yokoyama Y, Itoh M. Role of endogenous nitric oxide in ischaemia-reperfusion injury of rat gastric mucosa. J Gastroenterol Hepatol. 1998 Oct;13(10):997-1001. doi: 10.1111/j.1440-1746.1998.tb00560.x. PMID 9835314
- [Background] Bednar DA, Jain AK, Scott HJ. Mycotic abdominal aortic aneurysm: a case report. Can J Surg. 1985 Jan;28(1):23-4. PMID 3882200